CLINICAL TRIAL: NCT02323113
Title: An Open-Label, Phase 1b/2 Study Investigating Recommended Phase 2 Dose, Safety, Tolerability, and Preliminary Efficacy of TAK-659 in Adult Patients With Relapsed or Refractory Acute Myelogenous Leukemia (AML)
Brief Title: Safety, Tolerability, and Efficacy of TAK-659 in Adults With Relapsed or Refractory Acute Myelogenous Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business Decision; No Safety or Efficacy Concerns.
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C34002; U1111-1163-2185 (Registry Identifier: WHO)
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acute Myelogenous Leukemia
Keywords: Drug therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — TAK-659

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1b: TAK-659 (Experimental): TAK-659 tablets taken orally, once daily or twice daily on Days 1-28 in a 28 day cycle, for up to 12 cycles or until disease progression. Dosage of TAK-659 may increase in 20 mg increments using a 3 + 3 dose escalation design to determine a MTD and/or RP2D.
  Interventions: Drug: TAK-659
- Phase 2: TAK-659 (Experimental): TAK-659, tablets taken orally, once daily or twice daily on Days 1-28 in a 28 day cycle, for up to 12 cycles or until disease progression. Dosage for this phase will be determined from results of Phase 1b MTD/RP2D.
  Interventions: Drug: TAK-659

INTERVENTIONS:
Drug: TAK-659 — TAK-659 tablets.

SUMMARY:
The purpose of the Phase 1b dose finding phase is to determine the safety, tolerability, and maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of TAK-659 in participants with relapsed or refractory AML. The purpose of the Phase 2 expansion phase is to evaluate preliminary efficacy of TAK-659 in relapsed or refractory AML as measured by overall response rate (ORR).

DETAILED DESCRIPTION:
The drug being tested in this study is TAK-659. TAK-659 is being tested to treat people who have relapsed or refractory acute myelogenous leukemia (AML). This study will be conducted in 2 phases. The first phase will determine a safe and well-tolerated dose of TAK-659 to be used in the second phase, and the second phase will look at response to treatment in people who take TAK-659.

The study will enroll approximately 106 participants (approximately 40 in the first phase and 66 in the second phase). There will be two separate cohorts during Phase 2 portion of the study, one for participants with FLT-3 internal tandem duplication (ITD) mutations and the other for FLT-3 wild-type participants.

Phase 1b:

• TAK-659 60 milligram (mg) tablet starting dose escalated in 20 mg or higher increments to a maximum tolerated dose or RP2D

Phase 2:

• TAK-659 tablet at the maximum tolerated dose or RP2D determined in Phase 1b.

All participants will be asked to take their prescribed tablets at the same time each day throughout the study.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is up to 24 months (12 months of treatment and 12 months of follow up) unless the treating physician believes the participant would continue to derive benefit from the study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years or older.
2. Must have a histopathologically documented diagnosis of primary or secondary AML (excluding acute promyelocytic leukemia), as defined by World Health Organization (WHO) criteria (Jaffe et al, 2001), for whom no standard therapies are anticipated to result in a durable remission according to the clinical judgment of the principal investigator, or who refuses standard therapies (phase 1b and 2).
3. Participants for the phase 2 portion of the study must, in addition, meet the following:

   o Must be refractory to or relapsed after no more than 2 prior chemotherapy regimens. Re-induction with the same regimen or stem cell transplant will not be considered a separate regimen.
4. Eastern Cooperative Oncology Group performance status of 0 to 1.
5. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, or
   * Are surgically sterile, or
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 180 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together).

   Male participants, even if surgically sterilized (that is, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study treatment period and through 180 days after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods for the female partner], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception. Female and male condoms should not be used together).
6. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
7. In the absence of rapid progressive disease, the interval from prior systemic anticancer treatment to time of TAK-659 administration should be at least 2 weeks for cytotoxic agents (other than hydroxyurea), or at least 5 half-lives for noncytotoxic agents, and participants have to have recovered from acute toxicities of these therapies. Participants who are on hydroxyurea may be included in the study and may continue on hydroxyurea for the first 28 days while participating in this study.
8. Suitable venous access for the study-required blood sampling, including pharmacokinteic (PK) and pharmacodynamic (PD) sampling and blood transfusion support.
9. Clinical laboratory values as specified in the following:

   * Total bilirubin must be less than or equal to (<=) 1.5* the upper limit of normal (ULN).
   * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be less than or equal to (<=) 2.5*the ULN.
   * Lipase <=1.5*ULN and amylase <=1.5*ULN with no clinical symptoms suggestive of pancreatitis or cholecystitis.
   * Creatinine clearance greater than or equal to (>=) 60 milliliter per minute (mL/min) either as estimated by the Cockcroft-Gault equation or based on urine collection (12 or 24 hours).

Exclusion Criteria:

1. Clinically active central nervous system leukemia.
2. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 before first dose of study drug.
3. Any serious medical or psychiatric illness, including drug or alcohol abuse that could, in the investigator's opinion, potentially jeopardize the safety of the participant or interfere with the objectives of the study.
4. Systemic anti-cancer treatment (including investigational agents) <=21 days or <= 5*their half-lives before the first dose of study treatment. (For example, if the 5*the half-life is shorter than 21 days, 5*half-life should be used as the washout period. However, a minimum of 10 days should elapse from prior therapy to initiating protocol therapy).
5. Persistent clinically significant toxicity from prior chemotherapy that is Grade 2 or higher by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (v4.03).
6. Receipt of hematopoietic stem cell transplant (HSCT) within 60 days of the first dose of TAK-659; clinically significant graft-versus-host disease (GVHD) requiring ongoing immunosuppressive therapy post HSCT at the time of screening (use of topical steroids for ongoing skin GVHD is permitted).
7. Active, systemic infection requiring intravenous (IV) antibiotic, antifungal, or antiviral therapy or other serious infection within 14 days before the first dose of study drug.
8. Major surgery within 14 days before the first dose of study drug and have not recovered fully from any complications from surgery.
9. Radiotherapy less than 2 weeks before the first dose of study treatment or have not recovered from acute toxic effects from radiotherapy.
10. Known human immunodeficiency virus (HIV) positive (testing not required).
11. Known hepatitis B surface antigen-positive, known or suspected active hepatitis C infection (testing not required).
12. Evidence of currently uncontrolled cardiovascular conditions as listed in the protocol; acute myocardial infarction with 6 months before starting study drug; baseline QT interval (QTcF) greater than (>) 450 milliseconds (msec) (males) or > 475 msec (females); or abnormalities on baseline 12-lead electrocardiogram (ECG) that are considered clinically significant per investigator.
13. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of TAK-659 including difficulty swallowing tablets; diarrhea > Grade 1 despite supportive therapy.
14. Use or consumption of any of the following substances:

    * Medications or supplements that are known to be inhibitors of P-glycoprotein (P-gp) or strong inhibitors or inducers of Cytochrome (CY) P3A within 5 times the inhibitor half-life (if a reasonable half-life estimate is known) or within 7 days (if a reasonable half-life estimate is unknown) before the first dose of study drug. In general, the use of these agents is not permitted during the study except for AE management.
    * Medications or supplements that are known to be strong CYP3A mechanism based inhibitors or strong CYP3A inducers and/or P-gp inducers within 7 days or within 5 times the inhibitor or inducer half-life (whichever is longer) before the first dose of study drug. In general, the use of these agents is not permitted during the study except for AE management.
    * Grapefruit-containing food or beverages within 5 days before the first dose of study drug. Note that grapefruit-containing food and beverages are not permitted during the study.
15. White blood cell count > 50,000 per micro liter (/µL); hydroxyurea may be used to control the level of circulating leukemic blast cell counts prior to study entry and, if needed, concomitantly while on TAK-659 treatment during the first 28 days of the study. Hydroxyurea can be used up to a maximum dose of 5 gram per (g/) day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (17):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Oncology Specialists, S.C., Niles, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - North Shore Long Island Jewish Medical Center, New York, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - UC Health Clinical Trials Office, Cincinnati, Ohio
  - Baylor University Medical Center, Dallas, Texas
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Canada (3):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - Wake Forest University Baptist Medical Center, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Pratz KW, Kaplan J, Levy M, Bixby D, Burke PW, Erba H, Wise-Draper TM, Roboz GJ, Papadantonakis N, Rajkhowa T, Hernandez D, Dobler I, Gregory RC, Li C, Wang S, Stumpo K, Kannan K, Miao H, Levis M. A phase Ib trial of mivavotinib (TAK-659), a dual SYK/FLT3 inhibitor, in patients with relapsed/refractory acute myeloid leukemia. Haematologica. 2023 Mar 1;108(3):705-716. doi: 10.3324/haematol.2022.281216. PMID 36226495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 7 investigative sites in United States from 09 March 2015 to study end date:15 August 2018. An additional 8 sites were activated to participate in the Phase 2 expansion phase of the study, however, the Phase 2 portion of the study was not opened for enrollment.
Pre-assignment Details: Participants with relapsed or refractory acute myelogenous leukemia(AML)were enrolled in dose escalation phase of study to receive TAK-659 to determine maximum tolerated dose/recommended phase 2 dose. In dose expansion phase(Phase 2), participants refractory to or relapsed after <=2 prior chemotherapy regimens and with no prior exposure to any investigational FLT-3 inhibitors were to be enrolled, however, as per Sponsor's decision, the study terminated before initiation of the Phase 2.
Groups:
- TAK-659 60 mg QD: TAK-659, 60 mg tablets, orally, QD on Days 1 to 28 in each 28-day Cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 12 cycles.
- TAK-659 100 mg QD: TAK-659, 100 mg tablets, orally, QD on Days 1 to 28 in each 28-day Cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 12 cycles.
- TAK-659 120 mg QD: TAK-659, 120 mg, tablets, orally, QD on Days 1 to 28 in each 28-day Cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 12 cycles.
- TAK-659 140 mg QD: TAK-659, 140 mg, tablets, orally, QD on Days 1 to 28 in each 28-day Cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 12 cycles.
- TAK-659 160 mg QD: TAK-659, 160 mg, tablets, orally, QD on Days 1 to 28 in each 28-day Cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 12 cycles.
- TAK-659 60 mg BID: TAK-659, 60 mg, tablets, orally, BID on Days 1 to 28 in each 28-day Cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 12 cycles.
- TAK-659 80 mg BID: TAK-659, 80 mg tablets, orally, BID on Days 1 to 28 in each 28-day Cycle until disease progression or occurrence of unacceptable drug-related toxicities or discontinuation or up to 12 cycles.
- Phase 2 (Dose Expansion Phase): TAK-659 tablets at the maximum-tolerated dose (MTD)/recommended phase 2 dose (RP2D) determined from dose escalation phase, orally, QD or BID on Days 1 to 28 in each 28-day Cycle, for up to 12 cycles or until disease progression in participants who were to be entered in Phase 2.
Period: Overall Study
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID | Phase 2 (Dose Expansion Phase)
Started | 4 | 7 | 4 | 5 | 9 | 8 | 6 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 7 | 4 | 5 | 9 | 8 | 6 | 0
Not completed — Adverse Event | 3 | 3 | 2 | 5 | 8 | 3 | 6 | 0
Not completed — Progressive Disease | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Unsatisfactory Therapeutic Response | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Study Drug was Held due to AE for >21 Days, Therefore Participant was Discontinued Per Protocol | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID | Total
Number analyzed (Participants) | 4 | 7 | 4 | 5 | 9 | 8 | 6 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (19.62) | 59.3 (16.40) | 56.0 (18.89) | 60.0 (20.30) | 68.0 (7.35) | 50.3 (14.69) | 58.5 (13.98) | 59.4 (15.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 1 | 3 | 5 | 3 | 4 | 20
  Male | 4 | 3 | 3 | 2 | 4 | 5 | 2 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 3 | 7 | 4 | 5 | 9 | 6 | 6 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2 | 0 | 2 | 2 | 8
  White | 3 | 5 | 3 | 3 | 9 | 6 | 3 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 7 | 4 | 5 | 9 | 8 | 6 | 43
Height [Mean (Standard Deviation); unit: cm] — Population: Number of participants analyzed is the number of participants with data available for height at Baseline.
  cm
    number analyzed (Participants) | 4 | 5 | 4 | 5 | 9 | 8 | 6 | 41
    (all) | 166.9 (6.80) | 168.1 (15.15) | 169.2 (6.35) | 170.4 (15.06) | 168.8 (11.75) | 176.8 (10.29) | 169.6 (13.49) | 170.4 (11.49)
Weight [Mean (Standard Deviation); unit: kg] | 63.30 (10.692) | 77.16 (18.963) | 79.48 (13.133) | 75.62 (15.049) | 78.48 (27.515) | 90.41 (23.728) | 89.82 (24.609) | 80.41 (21.645)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) and Serious Adverse Event (SAE)
Description: AE meant any untoward medical occurrence in a participant or participant administered a pharmaceutical product; the untoward medical occurrence did not necessarily have a causal relationship with this treatment. SAE is any untoward medical occurrence that at any dose may result in death, life-threatening, required in participant hospitalization or prolongation of an existing hospitalization or can be a medically important event. TEAEs were defined as any AE that occurs after administration of the first dose of study treatment and up through 28 days after the last dose of study medication, or until the start of subsequent antineoplastic therapy, whichever occurs first.
Time Frame: From the first dose of study drug through 28 days after the last dose of study drug or until the start of subsequent antineoplastic therapy, whichever occurred first (Up to 13 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID
Number analyzed (Participants) | 4 | 7 | 4 | 5 | 9 | 8 | 6
Participants
  TEAEs | 4 | 7 | 4 | 5 | 9 | 8 | 6
  SAEs | 4 | 6 | 4 | 5 | 9 | 7 | 6

2. Primary Outcome: Phase 1b: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Toxicity was evaluated according to the NCI CTCAE, v4.03. DLT was defined as any of the following considered related to any of the treatment, by investigator: Prolonged myelosuppression with persistence of Grade ≥4 neutropenia or thrombocytopenia in absence of leukemia (blast count <5% in bone marrow) ≥42 days after initiation of Cycle 1 therapy; Any Grade ≥3 nonhematologic toxicity with exceptions- Grade 3 nausea or emesis resolved to Grade ≤1 or baseline in a week after use of optimal antiemetic regimen. Grade 3 diarrhea that resolved to Grade ≤1 or baseline in a week after receiving maximal supportive therapy, Brief (<1 week) Grade 3 fatigue, Asymptomatic Grade 3 laboratory abnormalities that were not clinically significant; Failure to administer ≥75% of planned doses of study drug due to TAK-659 -related or possibly related hematological or nonhematologic toxicities; related Grade ≥2 nonhematologic toxicities that required dose reduction or discontinuation of therapy.
Time Frame: Up to Cycle 1 (28 days)
Population: DLT-evaluable population include all participants in the phase 1b portion of the study at each dose cohort who either experienced a DLT during Cycle 1 or completed at least 75% of planned doses of TAK-659 and had sufficient follow-up data to allow both the sponsor and investigators to determine whether a DLT occurred.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 6 | 7 | 6
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 3

3. Primary Outcome: Phase 1b: Number of Participants With Clinically Significant Laboratory Findings Reported as TEAEs
Description: Clinical laboratory evaluations were performed locally for Hematology, Serum Chemistry, Urinalysis. Any abnormal laboratory values were reported as a TEAE if that value led to discontinuation or delay in treatment, dose modification, therapeutic intervention, or was considered by the investigator to be a clinically significant change from Baseline.
Time Frame: From first dose of study drug through 28 days after the last dose of study drug or until the start of subsequent antineoplastic therapy, whichever occurred first (Up to 13 months)
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID
Number analyzed (Participants) | 4 | 7 | 4 | 5 | 9 | 8 | 6
Participants
  Febrile neutropenia | 0 | 3 | 3 | 4 | 5 | 5 | 6
  Anaemia | 0 | 1 | 1 | 1 | 4 | 2 | 3
  Thrombocytopenia | 1 | 3 | 1 | 0 | 0 | 0 | 0
  Pancytopenia | 0 | 1 | 0 | 0 | 2 | 0 | 0
  Leukocytosis | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Leukopenia | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Neutropenia | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Thrombocytosis | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased | 0 | 5 | 2 | 3 | 5 | 3 | 4
  Amylase increased | 0 | 4 | 1 | 2 | 4 | 3 | 2
  Alanine aminotransferase increased | 0 | 3 | 2 | 2 | 3 | 1 | 3
  Lipase increased | 0 | 2 | 1 | 2 | 4 | 3 | 2
  Platelet count decreased | 0 | 0 | 0 | 1 | 3 | 1 | 4
  Blood lactate dehydrogenase increased | 1 | 1 | 0 | 2 | 1 | 0 | 2
  White blood cell count decreased | 0 | 0 | 0 | 0 | 2 | 3 | 2
  Neutrophil count decreased | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Gamma-glutamyltransferase increased | 1 | 0 | 1 | 1 | 1 | 1 | 0
  Blood alkaline phosphatase increased | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Blood creatinine increased | 0 | 1 | 1 | 0 | 0 | 1 | 1
  Blood calcium decreased | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Blood phosphorus decreased | 0 | 0 | 0 | 1 | 0 | 2 | 0
  Blood bilirubin increased | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Blood potassium decreased | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Blood uric acid increased | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Haemoglobin decreased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lymphocyte count increased | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Transaminases increased | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Hypophosphataemia | 1 | 1 | 2 | 1 | 2 | 0 | 4
  Hypocalcaemia | 0 | 0 | 1 | 4 | 1 | 1 | 2
  Hypokalaemia | 0 | 3 | 1 | 1 | 1 | 1 | 1
  Hypomagnesaemia | 1 | 1 | 1 | 3 | 0 | 0 | 1
  Hyperkalaemia | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Hyperuricaemia | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Hyponatraemia | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Hyperamylasaemia | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycaemia | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperlipasaemia | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatraemia | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperphosphataemia | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hypoglycaemia | 0 | 0 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Phase 1b: Number of Participants With Clinically Significant Vital Sign Findings Reported as TEAEs
Description: Vital signs measurement (blood pressure, heart rate, and temperature) were performed before dosing on visit days and as clinically indicated. Any vital sign finding were reported as a TEAE if that value led to discontinuation or delay in treatment, dose modification, therapeutic intervention, or was considered by the investigator to be a clinically significant change from Baseline.
Time Frame: as for outcome 3
Population: Safety population included all enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID
Number analyzed (Participants) | 4 | 7 | 4 | 5 | 9 | 8 | 6
Participants
  Weight Increased | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Tachycardia | 0 | 1 | 1 | 0 | 1 | 0 | 1
  Hypertension | 1 | 0 | 2 | 0 | 1 | 0 | 0
  Hypotension | 0 | 0 | 0 | 0 | 2 | 1 | 0
  Pyrexia | 1 | 2 | 1 | 1 | 4 | 0 | 2

5. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: ORR was defined as percentage of participants who achieved complete response (CR), complete response with incomplete platelet recovery (CRp), incomplete hematologic recovery (CRi), partial hematologic recovery (CRh), composite complete remission (CRc), and partial response (PR) in response-evaluable population. CR: morphologic leukemia-free state and have absolute neutrophil count (ANC) of more than 1000/μL and platelets of ≥100,000/μL. CRp: satisfied all CR criteria except platelets <100,000/μL. CRi: fulfill all of the criteria for CR after chemotherapy except for residual neutropenia (<1000/μL) or thrombocytopenia (<100,000/μL). CRh: no evidence of peripheral blasts and partial recovery of peripheral blast counts including ANC above 500/μL and platelets above 50,000/μL. CRc: sum of participant achieving CR, CRh, CRi, or CRp. PR required all of the hematologic values for a CR but with a decrease of at least 50% in the percentage of blasts to 5% to 25% in bone marrow aspirate.
Time Frame: Up to 13 months
Population: This outcome measure was not analyzed as the expansion phase 2 portion of the study was not opened for enrollment and the planned analyses were not conducted due to early termination of study.
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: DOR was defined as the time from the date of first documentation of a response to the date of first documented progressive disease (PD). PD was defined as >50% increase in bone marrow blasts from baseline value.
Time Frame: Up to 13 months
Population: as for outcome 5
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: TTP was defined as the time from the date of first study drug administration to the date of first documentation of PD by the investigator. PD was defined as >50% increase in bone marrow blasts from baseline value.
Time Frame: Up to 13 months
Population: This outcome measure was not analyzed as expansion phase 2 portion of the study was not opened for enrollment and planned analyses were not conducted due to early termination of study.
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase 2: Mortality Rate at Months 3 and 6
Description: Percentage of participants who died at Months 3 and 6.
Time Frame: Months 3 and 6
Population: This outcome measure was not analyzed as the expansion phase 2 portion of the study was not opened for enrollment and planned analyses were not conducted due to early termination of study.
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as the time from the date of study entry to the date of death.
Time Frame: Up to 13 months
Population: as for outcome 5
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

10. Secondary Outcome: Phase 2: Overall Response Rate (ORR) in FLT-3-internal Tandem Duplication (ITD) Mutant Versus Wild Type (WT) Populations
Description: as for outcome 5
Time Frame: Days 22 to 28 of Cycles 1, 2, 4 and 5 (each cycle was of 28-days)
Population: as for outcome 5
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase 2: Duration of Response (DOR) in FLT-3-ITD Mutant Versus WT Populations
Description: DOR was defined as the time from the date of first documentation of a response to the date of first documented PD. PD was defined as >50% increase in bone marrow blasts from baseline value.
Time Frame: Up to 13 months
Population: as for outcome 8
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase 2: Time to Progression (TTP) in FLT-3-ITD Mutant Versus WT Populations
Description: as for outcome 7
Time Frame: Up to 13 months
Population: as for outcome 8
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 2: Mortality Rate in FLT-3-ITD Mutant Versus WT Populations
Description: Number of participants who died at Months 3 and 6.
Time Frame: Months 3 and 6
Population: as for outcome 8
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase 2: Overall Survival (OS) in FLT-3-ITD Mutant Versus WT Populations
Description: OS was defined as the time from the date of study entry to the date of death.
Time Frame: Cycle 1 (28-day Cycle), Day 1 to 12 months
Population: as for outcome 7
Arm/Group | Phase 2 (Dose Expansion Phase)
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 1: Cmax: Maximum Observed Plasma Concentration After Single Dose (Day 1) and Multiple Dose (Day 15) for TAK-659
Time Frame: Cycle 1 (28-day cycle), Days 1 and 15 pre-dose and at multiple time points (Up to 24 hours for QD arms and Up to 8 hours for BID arms) post-dose
Population: PK-evaluable population included all participants in the acute myelogenous leukemia dose escalation cohorts who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID
Number analyzed (Participants) | 4 | 7 | 4 | 5 | 9 | 8 | 6
ng/mL
  Cycle 1 Day 1 | 74.39 (32.27) | 157.21 (41.54) | 211.32 (41.98) | 310.76 (30.13) | 322.32 (68.92) | 87.86 (96.10) | 122.59 (42.81)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 2 | 4 | 5 | 5 | 4
  Cycle 1 Day 15 | 188.48 (46.25) | 256.10 (44.58) | 213.13 (35.55) | 574.23 (25.98) | 404.07 (53.48) | 120.39 (60.27) | 299.01 (43.89)

16. Secondary Outcome: Phase 1: Tmax: Time to Reach the Maximum Observed Plasma Concentration After Single Dose (Day 1) and Multiple Dose (Day 15) for TAK-659
Time Frame: as for outcome 15
Population: as for outcome 15
Measure: Median (Full Range); unit: hrs
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID
Number analyzed (Participants) | 4 | 7 | 4 | 5 | 9 | 8 | 6
hrs
  Cycle 1 Day 1 | 2.41 [0.5 to 3.0] | 2.08 [0.8 to 3.0] | 2.53 [2.0 to 3.0] | 3.03 [1.0 to 3.1] | 1.17 [0.5 to 4.0] | 2.63 [0.5 to 3.8] | 2.08 [1.0 to 3.8]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 2 | 4 | 5 | 5 | 4
  Cycle 1 Day 15 | 1.97 [1.0 to 2.2] | 2.00 [1.9 to 3.1] | 2.10 [1.2 to 3.0] | 2.04 [1.0 to 4.0] | 2.97 [2.0 to 4.0] | 2.17 [1.0 to 4.1] | 1.48 [0.7 to 2.1]

17. Secondary Outcome: Phase 1: AUC0-24: Area Under the Plasma Concentration-Time Curve During a Dosing Interval After Single Dose (Day 1) and Once-Daily (QD) Multiple Dose (Day 15) for TAK-659
Description: AUC0-24 was analyzed in the QD arms/cohorts as their sampling was done up to 24 hours.
Time Frame: Cycle 1 (28-day cycle), Days 1 and 15 pre-dose and at multiple time points (Up to 24 hours for QD arms) post-dose
Population: Participants from PK-evaluable population included all participants in the acute myelogenous leukemia dose escalation cohorts who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters who received QD dosing of TAK-659. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD
Number analyzed (Participants) | 4 | 7 | 4 | 5 | 9
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 7 | 4 | 5 | 9
  Cycle 1 Day 1 | 796.8688 (29.8559) | 1244.4982 (32.8536) | 2072.1874 (55.3105) | 2563.5593 (21.0820) | 3188.8032 (59.6781)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 5 | 2 | 3 | 4
  Cycle 1 Day 15 | 1767.7607 (41.9029) | 2368.2318 (43.8496) | 2535.7901 (19.5210) | 4636.1667 (23.7653) | 4390.3805 (42.5850)

18. Secondary Outcome: Phase 1: AUC0-8: Area Under the Plasma Concentration-Time Curve During a Dosing Interval After Single Dose (Day 1) and Twice-Daily (BID) Multiple Dose (Day 15) for TAK-659
Description: AUC0-8 was analyzed in the BID arms/cohorts as their sampling was done up to 8 hours.
Time Frame: Cycle 1 (28-day cycle), Days 1 and 15 pre-dose and at multiple time points (Up to 8 hours for BID arms) post-dose
Population: Participants from PK-evaluable population included all participants in the acute myelogenous leukemia dose escalation cohorts who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters who received BID dosing of TAK-659. Number analyzed is number of participants with data available for analysis at the given time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | TAK-659 60 mg BID | TAK-659 80 mg BID
Number analyzed (Participants) | 8 | 6
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 7 | 6
  Cycle 1 Day 1 | 369.3765 (65.9672) | 519.9999 (44.9975)
  Cycle 1 Day 15: number analyzed (Participants) | 5 | 3
  Cycle 1 Day 15 | 718.2914 (47.5599) | 1239.4346 (31.9812)

19. Secondary Outcome: Phase 1: CL/Fss: Apparent Clearance After Extravascular Administration at Steady State After Once-Daily (QD) Multiple Dose (Day 15) for TAK-659
Time Frame: Cycle 1 (28-day cycle), Day 15 pre-dose and at multiple time points (Up to 24 hours for QD arms) post-dose
Population: PK-evaluable population included all participants in the acute myelogenous leukemia dose escalation cohorts who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Overall number analyzed is the number of participants with data available for analysis at the given timepoint. Only QD dosing Cohorts were analyzed for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD
Number analyzed (Participants) | 3 | 5 | 2 | 3 | 4
L/h | 33.9412 (41.9029) | 42.2256 (43.8496) | 47.3225 (19.5210) | 30.1974 (23.7653) | 36.4433 (42.5850)

20. Secondary Outcome: Phase 1: Rac(AUC0-24): Accumulation Ratio Based on AUC0-24 After Once-Daily (QD) Multiple Dose (Day 15) for TAK-659
Description: Accumulation ratio (based on AUC0-24), calculated as AUC0-24 after multiple dosing (at steady state)/AUC0-24 after a single dose.
Time Frame: Cycle 1 (28-day cycle), Day 15 pre-dose and at multiple time points (up to 24 hours for QD arms) post-dose
Population: Participants from PK-evaluable population included all participants in the acute myelogenous leukemia dose escalation cohorts who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters who received QD dosing of TAK-659. Overall number analyzed are the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD
Number analyzed (Participants) | 2 | 5 | 2 | 3 | 4
ratio | 2.7001 (20.7227) | 1.7936 (32.6687) | 1.5697 (11.4956) | 1.9398 (7.1129) | 2.0033 (28.3167)

21. Secondary Outcome: Phase 1: Rac(AUC0-8): Accumulation Ratio Based on AUC0-8 After Twice-Daily (BID) Multiple Dose (Day 15) for TAK-659
Description: Accumulation ratio (based on AUC0-8), calculated as AUC0-8 after multiple dosing (at steady state)/AUC0-8 after a single dose.
Time Frame: Cycle 1 (28-day cycle), Day 15 pre-dose and at multiple time points (up to 8 hours for BID arms) post-dose
Population: Participants from PK-evaluable population included all participants in the acute myelogenous leukemia dose escalation cohorts who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters who received BID dosing of TAK-659. Overall number analyzed are the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | TAK-659 60 mg BID | TAK-659 80 mg BID
Number analyzed (Participants) | 5 | 3
ratio | 2.3819 (45.4917) | 2.6371 (36.8694)

22. Secondary Outcome: Phase 1: PTR: Peak Trough Ratio After Multiple Dose (Day 15) for TAK-659
Description: The ratio of the maximum observed plasma concentration to the observed trough plasma concentration, where trough concentration is the concentration at the end of the dosing interval at steady-state before the next dose is administered.
Time Frame: Cycle 1 (28-day cycle), Day 15 pre-dose and at multiple time points (Up to 24 hours for QD arms and Up to 8 hours for BID arms) post-dose
Population: PK-evaluable population included all participants in the acute myelogenous leukemia dose escalation cohorts who had sufficient dosing and PK data to reliably estimate 1 or more PK parameters. Overall number analyzed are the number of participants with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID
Number analyzed (Participants) | 3 | 5 | 2 | 4 | 5 | 5 | 4
ratio | 4.8957 (21.1877) | 6.1564 (56.0024) | 4.1585 (24.0807) | 6.7852 (35.6808) | 4.7045 (24.8880) | 1.8886 (31.4783) | 2.6415 (27.6855)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 28 days after the last dose of study drug or until the start of subsequent antineoplastic therapy, whichever occurred first (Up to 13 months)
Description: At each visit the investigator had to document any occurrence of adverse events and clinically significant abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TAK-659 60 mg QD | TAK-659 100 mg QD | TAK-659 120 mg QD | TAK-659 140 mg QD | TAK-659 160 mg QD | TAK-659 60 mg BID | TAK-659 80 mg BID
All-Cause Mortality (participants affected / at risk) | 1/4 | 3/7 | 3/4 | 4/5 | 7/9 | 4/8 | 4/6
Serious Adverse Events (participants affected / at risk) | 4/4 | 6/7 | 4/4 | 5/5 | 9/9 | 7/8 | 6/6
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 4/4 | 5/5 | 9/9 | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-659 60 mg QD (N=4) | TAK-659 100 mg QD (N=7) | TAK-659 120 mg QD (N=4) | TAK-659 140 mg QD (N=5) | TAK-659 160 mg QD (N=9) | TAK-659 60 mg BID (N=8) | TAK-659 80 mg BID (N=6)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 3 | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungaemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fusarium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia escherichia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary mycosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 3 | 4 | 3 | 5
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 3 | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lactobacillus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-659 60 mg QD (N=4) | TAK-659 100 mg QD (N=7) | TAK-659 120 mg QD (N=4) | TAK-659 140 mg QD (N=5) | TAK-659 160 mg QD (N=9) | TAK-659 60 mg BID (N=8) | TAK-659 80 mg BID (N=6)
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 2 | 2 | 3 | 4 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 2 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral mucosa haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 5 | 2 | 3 | 5 | 3 | 4
Amylase increased (Investigations) | 0 | 4 | 1 | 2 | 4 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 3 | 2 | 2 | 3 | 1 | 3
Lipase increased (Investigations) | 0 | 2 | 1 | 2 | 4 | 3 | 2
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 3 | 1 | 4
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 2 | 1 | 0 | 2
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 3 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 1
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Human rhinovirus test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pseudomonas test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respirovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Streptococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urine output increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 4 | 2 | 0 | 3 | 3 | 1
Chills (General disorders) | 0 | 2 | 1 | 1 | 2 | 2 | 1
Pyrexia (General disorders) | 0 | 2 | 1 | 1 | 3 | 0 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 1
Pain (General disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Unevaluable event (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 2 | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4 | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 1 | 1 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperamylasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 4 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 1 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1 | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 4 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 2 | 0 | 3 | 4 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 1 | 4 | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypogeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 2 | 3 | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 4 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2 | 1 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Splenic lesion (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scleral hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scleral oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Acinetobacter bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2 | 2 | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental fatigue (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Testicular oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT02323113/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT02323113/SAP_001.pdf